CLINICAL TRIAL: NCT02300584
Title: Distance Savvy: Testing Tele-Savvy, a Distance Dementia Family Caregiver Education Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Kenneth Hepburn, Kenneth Hepburn PhD, Emory University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00074715
Record Dates: First submitted 2014-11-21; First posted 2014-11-25 (Estimated); Last update posted 2016-09-08 (Estimated); Status verified 2016-09

CONDITIONS: Dementia; Alzheimer's Disease; Depression
MeSH Terms: conditions — Dementia; Alzheimer Disease; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Prototype Program (Experimental): The Savvy Caregiver (Savvy) - program delivered on an iPad (a tablet computer with an internet connection) extends over a six week period. Caregivers are asked to view brief daily videos (8-12 minutes) on the iPad. Once each week, a group of caregivers joins in a videoconference (an hour) with one or two trained leaders to review material from the week and to learn new material.
  Interventions: Behavioral: Tele-Savvy; Other: iPad
- Field Program (Experimental): The Savvy Caregiver (Savvy) - program delivered on an iPad (a tablet computer with an internet connection) extends over a six week period. Caregivers are asked to view brief daily videos (8-12 minutes) on the iPad. Based on the feedback from the prototype program, the videos may vary. Once each week, a group of caregivers joins in a videoconference (an hour) with one or two trained leaders to review material from the week and to learn new material.
  Interventions: Behavioral: Tele-Savvy; Other: iPad

INTERVENTIONS:
Behavioral: Tele-Savvy — as a program delivered on an iPad with daily instructional video segments (8-12 minutes each)
  Arms: Prototype Program
Behavioral: Tele-Savvy — as a program delivered on an iPad with daily instructional video segments (8-12 minutes each). Videos may be modified after feedback from Prototype arm.
  Arms: Field Program
Other: iPad — a tablet computer with an internet connection

SUMMARY:
The purpose of this study is to refine and test the web-based delivery of a well-established in-person group program that provides information and education to informal caregivers (family and friends) of persons with Alzheimer's disease (or related illnesses).

DETAILED DESCRIPTION:
The pilot project proposed will allow the investigators to use telehealth methods to deliver the Savvy Caregiver, an evidence-based dementia caregiver psychoeducation program, to family caregivers of community-dwelling persons with dementing illnesses (PWD) for whom attending in-person meetings poses difficulties. The program - named Tele-Savvy - uses iPad and PC technology and on-line conferencing capacity to deliver the program through daily asynchronous self-learning modules and weekly, hour-long synchronous group meetings with program facilitators. Tele-Savvy addresses all of the learning objectives of the current in-person Savvy program (Savvy entails in-person participation in six weekly two-hour group sessions).

ELIGIBILITY:
Inclusion Criteria:

* an informal caregiver for a person with a dementing disorder, such as Alzheimer's disease
* able to speak, read, and understand English
* has access to a computer with internet connection
* lives in the US

Exclusion Criteria:

* unwilling to participate in data gathering

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2014-11; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
The number of participants who use at least half of the opportunities (half of the conferences and half of the daily lessons) | 6 weeks

SECONDARY OUTCOMES:
Change in Zarit Burden Interview Score | Baseline, 6 weeks
  A 22-item questionnaire in which subjects rate how often they experience negative feelings associated with caregiving. Each item rated on a 5 point scale anchored at 0 for "never" and 4 for "nearly always." Scores range from 0-88 with higher scores indicating increased burden of care.
Change in Center for Epidemiological Studies-Depression Scale Score | Baseline, 6 weeks
  A 20-item scale measuring general depression. Scores range from 0-60, with higher scores indicating greater general depression.
Change in State Trait Anxiety Index (STAI) Score | Baseline, 6 weeks
  State Trait Anxiety Index questionnaire consists of 40 questions with 20 items allocated to each of the State Anxiety and Trait Anxiety subscales. The scores for each subtest range from 20 to 80, with higher scores indicating higher levels of anxiety.
Change in Connor Davidson Resilience Scale (CD-RISC) | Baseline, 6 weeks
  The Connor-Davidson Resilience scale (CD-RISC) comprises of 25 items, each rated on a 5-point scale. A score of 0 is suggestive of no resilience, a score of 100 is suggestive of high level of resilience.
Change in Perceived Stress Scale | Baseline, 6 weeks
  The Perceived Stress Scale is a 10-item questionnaire, on a 4-point scale (0 = Never, 4 = Very Often). Scores range from 0-40, with higher scores reflecting greater perceived stress.
Change in Caregiver Self-Efficacy Score | Baseline, 6 weeks
  Caregiver self-efficacy was measured by the Revised Checklist for Caregiving Self-Efficacy; the scale consists of 17 items which are rated from 0 - 100% confidence. The total score is summed from these percentages and ranges from 0 - 1700 where higher scores indicate a higher level of confidence.
Change in Personal Mastery scale | Baseline, 6 weeks
  Personal Mastery scale is a seven item, five-point Likert scale. Scoring is done by summing item scores for a total score (possible range 7-35) with higher scores indicating higher levels of mastery.
Change in Revised Memory and Behavior Problem Checklist | Baseline, 6 weeks
  This scale measures the type/number of dementia patients disturbing behaviors, and how much they bother caregivers with 24 items describing possible troublesome behaviors that the patient might evidence in the past month. Caregivers are first asked whether the dementia patient had displayed any of these in the time period, and secondly to rate on a 5-point scale (0=not at all; 4= extremely) how much this "bothered or upset" them. A "conditional bother" score is calculated which is the "upset" or "bother" ratings for only the problematic behavior that occurred. The scale refers to the caregiver. Minimum score (best value)=0. Maximum score (worst value)=4. Higher values represent a worse outcome.
Change in Lawton Activities of Daily Living (ADL) / Instrumental Activities of Daily Living (IADL) Scale | Baseline, 6 weeks
  Lawton ADL/IADL is caregiver reported performance of personal and instrumental activities of daily living (ADLs). There are 6 personal ADLs (i.e. dressing, grooming, eating, etc) and 8 instrumental ADLs (i.e. managing finances, transportation, food preparation) which are assessed. Each item is awarded 2 points for fully independent, 1 point for minimal or moderate support required, and 0 points for full support. Maximum score for independence with all personal and instrumental ADL's is 28.

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Hepburn, Ph.D., Principal Investigator — Emory University
Locations (1):
- Emory Alzheimer's Disease Research Center, Atlanta, Georgia, United States